Study Title: A Pilot Study Investigating the nCAP Signal Relief Patch in Subjects Undergoing Primary Hip or Knee Replacement Surgery – A Pilot Trial

Principal Investigator: Jacques E. Chelly, MD, PhD, MBA

IRB: STUDY22010018 NCT: 05252858

Statistical Analysis Plan Approval Date: 02/01/2022

Power calculation is for an anticipated 60 subjects who underwent TKA. Data is to be analyzed using intend-to-treat analysis plan. Data collection in this study includes the following measurements:

- Total opioid consumption (OME mg),
- Pain at rest and during movement rated on a standard Numerical Rating Scale (NRS, 0 = no pain and 10 = the worst pain imaginable),
- Area under the curve (AUC) for pain scores collected on POD 1, 2, 3, 7, 14, and 30,
- Time to discharge from the recovery room,
- Time to discharge from the hospital, and
- Overall subject satisfaction at the time of hospital discharge

The number of subjects requesting a prescription refill during the first 30-days post-operative will be calculated using the Pennsylvania Data Management Program.

Student's t-test, non-parametric Kruskal-Wallis test, or Pearson's chi-square test were used to determine differences in the distribution of continuous outcomes, and the chi-square test or exact test was used for differences in proportions for categorical outcomes between the treatment and placebo arms. Data will be presented as mean  $\pm$  standard deviation (SD) with a standard alpha set at 0.05.